CLINICAL TRIAL: NCT06223880
Title: A Randomized, Double-blind, Active-controlled Study of AXS-05 for the Prevention of Relapse of Depressive Symptoms
Brief Title: A Study to Evaluate the Efficacy of AXS-05 Compared to Bupropion in Preventing the Relapse of Depressive Symptoms
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AXS-05-MDD-401
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder
Keywords: AXS-05; Dextromethorphan; Bupropion; MDD; Depression; Relapse of depressive symptoms; NMDA receptor antagonist; Sigma-1 receptor agonist; Norepinephrine reuptake inhibitor; Dopamine reuptake inhibitor; Axsome Therapeutics
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-05 (Experimental): AXS-05 tablets, taken twice daily
  Interventions: Drug: AXS-05
- Bupropion (Active Comparator): Bupropion tablets, taken twice daily
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: AXS-05 — Up to 10 weeks in open-label period;
  Up to 26 weeks in double-blind period
  Arms: AXS-05
Drug: Bupropion — Up to 26 weeks in double-blind period
  Arms: Bupropion

SUMMARY:
This is a randomized, double-blind, active-controlled, multi-center study to evaluate the efficacy of AXS-05, compared to bupropion, in preventing the relapse of depressive symptoms in subjects with major depressive disorder (MDD) who have responded to treatment with AXS-05.

DETAILED DESCRIPTION:
Eligible subjects will receive open-label AXS-05 during the 10-week open-label treatment period, during which they will be monitored for response and remission. Subjects meeting the response and remission criteria during the open-label period will be randomized (1:1) to the double-blind period to continue treatment with AXS-05 or switch to treatment with bupropion (105 mg) tablets. Randomized subjects will receive double-blind treatment for 26 weeks or until they experience a relapse.

ELIGIBILITY:
Inclusion Criteria:

* Currently meets DSM-5 criteria for diagnosis of MDD without psychotic features
* Current major depressive episode of at least 4 weeks in duration

Exclusion Criteria:

* Previously participated in another clinical study of AXS-05; received any investigational drug or device treatment within 30 days of (Screening) Visit 1, or has been prescribed Auvelity.
* Unable to comply with study procedures
* Medically inappropriate for study participation in the opinion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to relapse of depressive symptoms | up to 26 weeks

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Clinical Research Site, Bellflower, California
  - Clinical Research Site, Lafayette, California
  - Clinical Research Site, Oceanside, California
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, Riverside, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Upland, California
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Doral, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Chicago, Illinois
  - Clinical Research Site, Overland Park, Kansas
  - Clinical Research Site, New Orleans, Louisiana
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Saint Charles, Missouri
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Cherry Hill, New Jersey
  - Clinical Research Site, Toms River, New Jersey
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, Mount Kisco, New York
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Edmond, Oklahoma
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, Friendswood, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Wichita Falls, Texas
  - Clinical Research Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com